CLINICAL TRIAL: NCT06560840
Title: Effectiveness of Gut Microbiota-targeted Diatery Intervention in Preventing Atherosclerotic Cardiovascular Disease Among Older People Living With HIV
Brief Title: Effectiveness of Gut Microbiota-targeted Diatery Intervention Among Older People Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junwen Yu, PhD candidate, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SZ-2024-008
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hiv; Atherosclerosis; Diet, Healthy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Atherosclerosis | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive the gut microbiota targeted dietary intervention thrice weekly for 3 months, accompanied by bi-weekly healthy diet guidance for the same duration. The intervention will span three months, followed by a three-month follow up period
  Interventions: Other: dietary intervention
- control group (No Intervention): The control group will continue routine follow-up and health education practices.

INTERVENTIONS:
Other: dietary intervention — The dietary intervention targeted at gut microbiota. Each participant's dietary habits,food preferences and economic level were taken into account. The dietary intervention was delivered by sending meals. To ensure the freshness and quality of the ingredients, 2 dedicated researchers were jointly responsible for the procurement of fresh ingredients, which were purchased through regular channels on Monday, Wednesday and Friday mornings. Meals will be delivered three times a week for a 12-week intervention period. Guided dietary follow-up was conducted through WeChat or telephone follow-up. The researcher will provide cooking instruction or dietary pattern guidance every two weeks.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to conduct a dietary intervention targeting HIV specific gut microbiota alterations for primary atherosclerotic cardiovascular disease (ASCVD) prevention and evaluate its effectiveness in preventing ASCVD among older people living with HIV (PLWH).

DETAILED DESCRIPTION:
The investigators utilize a pragmatic randomized controlled trial design to evaluate the effectiveness of dietary intervention in real-world conditions, without strict control, thereby enhancing the generalizability and clinical applicability of our study findings. Participants at Shenzhen Third People's Hospital, exhibiting HIV with CVD risk will be enrolled. Upon providing informed consent, participants will undergo dynamic randomization into intervention and control groups, aiming for a 1:1 ratio while preserving maximum unpredictability. The intervention group will receive the gut microbiota-targeted dietary intervention thrice weekly for 3 months, accompanied by bi-weekly healthy diet guidance for the same duration. Meanwhile, the control group will continue routine follow-up and health education practices. The intervention will span three months, followed by a three-month follow-up period. Data collection will occur at baseline, 3 months, and 6 months. Primary outcomes will assess ASCVD risk via the pooled cohort equation and evaluate gut microbiota diversity and composition. Secondary outcomes will encompass biomarkers and predictors associated with atherosclerotic cardiovascular disease, as well as symptoms related to the condition.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected patients diagnosed according to the diagnostic criteria of China AIDS diagnosis and treatment guidelines;
2. Aged 40 years and above;
3. at risk of CVD: having any two of those risk factors: dyslipidemia, DM or elevated blood glucose, smoking, hypertention or elevated blood pressure, metabolic syndrome,overweight/obesity; or PCE score>5%,
4. Those with a predicted survival time of >1 year;
5. No plans to leave the depth in the next 3 months;
6. Voluntary participation in this study and signing the informed consent

Exclusion Criteria:

1. Those with a previous history of CVD;
2. Those with HIV-related neurocognitive impairment, Alzheimer's disease or dementia, and a variety of serious opportunistic infections;
3. Currently suffering from malignant tumors, gastrointestinal diseases; People with an aversion to eating;
4. Allergic to nuts and fish;
5. People who take medicinal calcium >1000 mg per day or omega-3 supplements;
6. Plan to become pregnant within 6 months;
7. Are participating in other HIV-related or dietary intervention-related scientific research programs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
10-year ASCVD risk assessed by the Pooled Cohort Equations | baseline, 3-month and 6-month
  The Pooled Cohort Equations (PCE) will be utilized to estimate the 10-year risk of ASCVD. The required data will include age, gender, race, total cholesterol, HDL cholesterol, systolic blood pressure, hypertension treatment status, smoking status, and diabetes status. The PCE is a well-established and validated model for predicting ASCVD risk.
Gut microbiota diversity and composition | baseline and 3-month
  Fecal samples will be collected from study participants, and the diversity and composition of gut microbiota will be analyzed using 16S rRNA technology. Diversity Analysis: Bacterial richness and phylogenetic diversity within samples will be assessed using Faith's Phylogenetic Diversity and richness metrics. Taxonomic Composition: Relative abundance of specific bacterial taxa will be determined.

SECONDARY OUTCOMES:
Blood lipids | baseline and 3-month; 6-month only collect HDL-C, LDL-C, TC, and TG
  HDL-C, LDL-C, TC, TG, ApoA1, ApoB, Lp(a), and CR
Blood pressure | baseline, 3-month and 6-month
  Using the Omron automatic blood pressure monitor. Record the values displayed on the monitor for both systolic and diastolic pressures (mmHg). Repeat this process three times with a short rest period between each measurement, and calculate the average of the three readings for accurate results.
BMI | baseline, 3-month and 6-month
  To calculate BMI, the weight in kilograms is divided by the square of the height in meters (BMI = weight(kg) / height(m^2).
Waistline | baseline, 3-month and 6-month
  The measuring position is at the midpoint of the line between the anterior superior iliac ridge and the lower margin of the 12th rib. The tape is pressed against the skin, but it cannot be compressed.
ASCVD related symptoms | baseline, 3-month and 6-month
  Use the ACS symptom checklist and Memorial symptom assessment scale-heart failure to estimate ASCVD-related symptoms. The ACS Symptom Checklist is a validated instrument comprising 13 items designed to assess symptoms associated with ACS. Participants are asked to indicate whether each symptom is present (1) or absent (0). Each symptom is analyzed individually, and there is no composite score. The Memorial Symptom Assessment Scale-Heart Failure comprises 32 items, categorized into three subscales: physiological symptoms (n=21), psychological symptoms (n=6), and heart failure symptoms (n=5).
Three-day dietary diary | baseline, 3-month and 6-month
  Write down the food and drink the participants have in two working days and one rest day.
SF-36 Abbreviated Quality of Life Scale | baseline, 3-month and 6-month
  The scale was developed by the Boston Health Research Institute, based on the Rand Corporation Health Insurance project, to assess the degree of health change in the past year. In 1996, the International Quality of Life Evaluation Organization recommended the use of SF-36 for quality of life measurement. There are 36 items in the scale, of which item 2 is self-reported health change and does not participate in the score calculation of the scale. The remaining 35 entries are divided into eight dimensions, Including physical functioning, role-physical, bodily pain, and general health perceptions, vitality, social functioning, role-emotional, and mental health.
Physical activity assessed by IPAQ | baseline, 3-month and 6-month
  The international physical activity questionnaire (IPAQ) is a standardized tool for assessing an individual's physical activity level, originally developed by international organizations such as the World Health Organization and the U.S. Centers for Disease Control and Prevention. Available in short and long versions, it has been validated in more than 12 countries. The short version of the IPAQ consists of seven questions that assess an individual's level of physical activity by calculating total energy expended per week (MET-minutes/week).
Renal function index | baseline, 3-month and 6-month
  Cr and BUN
Liver function index | baseline, 3-month and 6-month
  total protein, albumin, globulin, white/ball ratio, total bilirubin, directly bound bilirubin, indirect bilirubin, total bile acid, alanine aminotransferase, aspartate aminotransferase, AST/ALT, and gamma-glutamyltransferase
Glucose | baseline, 3-month and 6-month
  Measurement of blood glucose levels
Inflammatory markers | baseline, 3-month
  IL-6, IL-8, TNF-a
HIV specific ASCVD risk factors | baseline, 3-month and 6-month
  HIV RNA, CD4 count, CD8 count
Dietary Regimen Adherence Scale | baseline, 3-month and 6-month
  Adapted from the 14-item Mediterranean diet adherence screener (MEDAS), which contains two questions about eating habits and eight questions about the frequency of consumption of typical foods in this dietary regimen, And 4 questions about foods not recommended in this diet. Each question is scored on the scale of compliance (1) or non compliance (0)
Food frequency questionnaire | baseline, 3-month
  Food frequency Questionnaire (FFQ 146) is from the complete food frequency questionnaire used by the National Institute of Nutrition and Food Safety of the Chinese Center for Disease Control and Prevention in a dietary survey in Beijing Exhibition Road community, including 146 food items

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Dr, Study Director — Shenzhen Third People's Hospital
Locations (1):
- The Third People's Hospital of Shenzhen, Shenzhen, China